CLINICAL TRIAL: NCT07394660
Title: The Effect of Remote Reiki Treatment on Hopelessness, Fatigue and Pain in Patients Awaiting Organ Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Ozlem Sahin Akboga, Assistant professor, Bozok University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BozokUnıversity; the author himself (Other: the author himself)
Record Dates: First submitted 2025-12-04; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Organ or Tissue Transplant; Complications; Reiki
Keywords: reiki; organ transplant; nursing; pain; Hopelessness
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This study is planned to be conducted as a randomized controlled trial with two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Experimental): remote reiki
  Interventions: Behavioral: remote reiki
- 2 (No Intervention): control

INTERVENTIONS:
Behavioral: remote reiki — Patients in the intervention group will be contacted by telephone. They will be provided with a suitable environment. A certified assistant researcher will initiate the remote Reiki application. Each application is expected to last an average of 35-40 minutes. The first remote Reiki session will be conducted on the evening of the patient's haemodialysis day. The sessions will take place three times a week for a total of four weeks. After the application is completed, vital signs will be taken again from the intervention group patients, and the Beck Hopelessness Scale, Fatigue Severity Scale, and Brief Pain Inventory will be completed. The data collection tool will be completed a second time the day after the last application and a third time one month later. The effects of Reiki therapy on hopelessness, fatigue, and pain will be evaluated using the Personal Information Form, Beck Hopelessness Scale, Fatigue Severity Scale, and Brief Pain Inventory.
  Arms: 1

SUMMARY:
The treatment and care of chronic kidney failure is a long-term process, and patients are significantly affected by this condition. The fact that patients spend much of their daily lives attending hemodialysis sessions two or three times a week considerably limits their life activities. dition to medical treatment, a non-pharmacological Therefore, individuals may become partially or completely dependent. Coping with various symptoms brought on by this chronic disease, adapting to the restrictions required by treatment, preventing complications, and improving quality of life also bring about physical, cognitive, and psychological challenges. Patients are aware that they can only regain their previous health through organ transplantation; however, since it is uncertain when a suitable donor will be found, they may experience intense feelings of hopelessness. The chronic illness itself and the hemodialysis sessions frequently lead to symptoms such as pain and fatigue. In admethod such as distant Reiki may be supportive in coping with symptoms like hopelessness, fatigue, and pain. Numerous evidence-based studies in the literature have demonstrated that distant Reiki practices support symptom management in many chronic diseases through their effects on the parasympathetic nervous system. However, the effects of distant Reiki on hopelessness, fatigue, and pain in individuals awaiting organ donation have not yet been investigated.

DETAILED DESCRIPTION:
Therefore, this study is planned to be conducted as a randomized controlled trial with two groups. Fifty patients awaiting organ donation who meet the inclusion criteria will be included in the study. Data will be collected using the "Personal Information Form," "Beck Hopelessness Scale," "Fatigue Severity Scale," and "Brief Pain Inventory." Analyses will be performed using an appropriate statistical software package. We believe that distant Reiki practices may have positive effects on hopelessness, fatigue, and pain among hemodialysis patients awaiting organ donation. It is known that the majority of nurses worldwide hold Reiki practice certifications and use this method in chronic diseases. The main aim of this study is to support symptom management and strengthen coping mechanisms in individuals through distant Reiki practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been undergoing haemodialysis for ≥ 6 months,
* Aged 18 years or older,
* Patients with chronic kidney disease,
* Can speak and understand Turkish and,
* Have a mobile phone and can use it will be included in the study.

Exclusion Criteria:

* Patients using psychotropic medication will not be included in the study.
* Patients who are unable to attend regular sessions will be excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-07-10 (Actual); Primary Completion 2025-08-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Hopelessness Level | From enrollment to the end of treatment at 8 weeks
  Hopelessness level will be assessed using the Beck Hopelessness Scale (BHS). The scale consists of 20 items and measures negative expectations about the future. Higher total scores indicate greater levels of hopelessness. Total scale score (0-20) Unit of Measure: Scale total score (0-20)
Pain Intensity and Pain Interference | From enrollment to the end of treatment at 8 weeks
  Pain intensity and pain-related interference with daily activities will be assessed using the numeric raito scale (NRS). The instrument evaluates pain severity and its impact on functioning. Pain severity score and pain interference score Unit of Measure: Scale total score (0-10)
Fatigue Severity | Baseline (first dialysis day), at 4 weeks (end of intervention), and 1 month after the final intervention session
  Fatigue severity will be measured using the Fatigue Severity Scale (FSS), a 9-item self-report questionnaire evaluating the impact of fatigue on daily functioning. Higher scores indicate greater fatigue severity.
  Unit of Measure: Total scale score (1-7)

SECONDARY OUTCOMES:
Systolic Blood Pressure | Baseline to 8 weeks
  Description:
  Systolic blood pressure measured under standardized resting conditions using an automated monitor.
  Unit of Measure: mmHg
Diastolic Blood Pressure | Baseline to 8 weeks
  Description:
  Diastolic blood pressure measured under standardized resting conditions using an automated monitor.
  Unit of Measure: mmHg
Heart Rate | Baseline to 8 weeks
  Description:
  Resting heart rate measured using an automated vital signs monitor. Unit of Measure: beats per minute (bpm)
Body Temperature | Baseline to 8 weeks
  Description:
  Body temperature measured using a digital thermometer under standardized conditions.
  Unit of Measure: °C

CONTACTS AND LOCATIONS:
Locations (1):
- Gökmedrese Dialasis Center, Yozgat, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results reported in publications (including outcome measure data, demographic variables, and relevant clinical variables) will be made available upon reasonable request to the corresponding author. All shared data will be fully anonymized to protect participant confidentiality and will exclude any personally identifiable information.
Supporting Information: SAP, CSR
Time Frame: Beginning 6 months after publication of the primary study results and up to 5 years following publication of the primary study results
Access Criteria: Researchers who provide a methodologically sound proposal and a reasonable scientific justification will be eligible to access the data. Requests should be submitted to the corresponding author via email. Data access may require approval by the principal investigator and the institutional ethics committee, where applicable. A data use agreement may be required prior to data sharing. Data will be available following publication of the primary study results and for a limited period thereafter.

REFERENCES:
- [Background] Akpinar, N. B., Unal, N., Alıncak, G., Pörücü, C., Yurtsever, S., & Karadurmus, N. (2025). The Power of Reiki: Its Effects on Pain and Biochemical Parameters in Patients Undergoing Bone Marrow Transplantation: A Randomized Prospective Controlled Study. Pain Management Nursing, 26(1), e24-e30.